CLINICAL TRIAL: NCT06762158
Title: Neoadjuvant Chemoradiotherapy Combined With Sequential Perioperative PD-1 Inhibitor for Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: NCRT Combined With Sequential Perioperative PD-1 Inhibitor for LAESCC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY2024-217-A
Record Dates: First submitted 2024-12-22; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: esophageal squamous cell cancer; neoadjuvant chemoradiotherapy; perioperative immunotherapy; PD-1 inhibitor
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Neoadjuvant Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perioperative toripalimab (Experimental): neoadjuvant chemoradiotherapy and perioperative toripalimab
  Interventions: Radiation: Neoadjuvant Chemoradiotherapy; Drug: neoadjuvant immunotherapy; Procedure: Surgery; Drug: adjuvant immunotherapy

INTERVENTIONS:
Radiation: Neoadjuvant Chemoradiotherapy — Neoadjuvant chemoradiotherapy:
  1. Radiation dose: 1.8Gy/Fx, DT41.4Gy/23Fx.
  2. Concurrent chemotherapy: Albumin-bound paclitaxel 60mg/m² + Cisplatin 25mg/m² on D1, D8, D15, D22, D29.
Drug: neoadjuvant immunotherapy — Begins on the second day after the completion of concurrent chemoradiotherapy, and no later than one week. Toripalimab 240mg Q3W, for a total of two cycles.
Procedure: Surgery — Preoperative assessment is conducted 3 weeks after the last neoadjuvant immunotherapy, and surgery is performed within 4-6 weeks. All patients undergo minimally invasive radical esophagectomy, either McKeown or Ivor-Lewis, with extended two-field or three-field lymph node dissection.
Drug: adjuvant immunotherapy — Whether to undergo postoperative adjuvant immunotherapy is determined based on the pathological response. Patients with pCR are only observed without receiving adjuvant treatment, while those not reaching pCR receive one year of adjuvant Toripalimab.

SUMMARY:
This study aims to examine the efficacy of the combination of neoadjuvant chemoradiotherapy and perioperative PD-1 inhibitor in patients with locally advanced esophageal squamous cell cancer and explore the predictive biomarkers for this regimen.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* Histologically or cytologically confirmed esophageal squamous cell cancer
* Stage T3-4aN0M0 or TanyN1-3M0 according to the American Joint Committee on Cancer staging manual eighth edition
* Eastern Cooperative Oncology Group performance status of 0 or 1
* he indexes of hematology, biochemistry and organ function meet the following requirements: a. white blood cell count (WBC) ≥ 3.0×109/L；b. neutrophil count (ANC) ≥ 1.5×109/L; c. platelets ≥ 85×109/L; d. hemoglobin ≥ 90g/L; e. total bilirubin ≤ 1.5 ULN; f. ALT ≤ 1.5 ULN; g. creatinine clearance rate >60 mL/min;
* The cardiopulmonary function needs to meet the following criteria: EF ≥ 55%, VC > 60%, FEV1 > 1.2L, FEV1%> 40%, DLco > 40%
* Women of childbearing age must undergo a pregnancy test within 7 days before enrollment for treatment, and only those with a negative result can be enrolled
* Voluntarily participating in this study

Exclusion Criteria:

* Patients with active infection within 2 weeks before the first use of the study drug
* A history of interstitial lung disease or non-infectious pneumonia
* A history of autoimmune diseases or abnormal immune system
* Patients who cannot tolerate chemoradiotherapy or surgery due to severe cardiac, lung dysfunction
* Patients diagnosed with any other malignant tumor within 5 years before enrollment, except for malignant tumors with low risk of recurrence and risk of death, such as fully treated basal cell or squamous cell skin and carcinoma in situ of the cervix;
* Known or suspected allergy or hypersensitivity to monoclonal antibodies, any ingredients of Toripalimab, and the chemotherapeutic drugs nab-paclitaxel or cisplatin
* A history of immunodeficiency，including a positive HIV test result or other acquired or congenital immunodeficiency diseases, a history of organ transplantation or allogeneic bone marrow transplantation
* Women during pregnancy or lactation
* Other situations not suitable for enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
pathologically complete response(pCR) | From date of surgery to 4 weeks later
  absence of viable tumor cells in the resected cancer specimen（ypT0N0）

SECONDARY OUTCOMES:
event free survival | 24 months
  From date of treatment until the date of death from any cause or the date of disease progression, assessed up to 24 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Radiation Oncology Department, Ren Ji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China